CLINICAL TRIAL: NCT03528655
Title: Influence of Decision Aids on the Choice of Mother-infant Rooming-in or Separation Care for Pregnant Women : a Randomized Controlled Trial
Brief Title: Influence of Decision Aids on the Choice of Mother-infant Rooming-in or Separation Care for Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Principal Investigator, Ka-Wai Tam, Director of Shared Decision Making Resource Center, Taipei Medical University Shuang Ho Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: N201802060
Record Dates: First submitted 2018-04-27; First posted 2018-05-18 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Pregnancy Related
Keywords: separation care; rooming-in care; patient decision aid
MeSH Terms: interventions — Decision Support Techniques

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Decision aid group (Experimental): Shared decision making using decision aid
  Interventions: Other: Decision aid
- Controlled group (No Intervention): Standard oral explanation with booklet.

INTERVENTIONS:
Other: Decision aid — Decision aid is a tool that helps pregnant women become involved in decision making on choosing rooming-in or separation care. Decision aid provides information about the options and outcomes, and by clarifying personal values.
  Arms: Decision aid group

SUMMARY:
During early postpartum period, mother-infant proximity is important for breastfeeding success. Rooming-in and separate care are both traditional practices. Rooming-in involves keeping the mother and the baby together in the same room after birth during hospitalization, whereas separate care keeps the baby in the hospital baby room. Shared decision making with decision aid (DA) is a way to provide information to pregnant women and to involve them in making decisions about their strategy on baby care. We have developed a DA to be administered during consultation for pregnant women, and conducted a randomized controlled trial (RCT) to evaluate the benefit of DA on decision making. The measurements include a battery of interview-based questionnaires and evaluations of decision regret. We expect the DA would benefit the intervention group in the aspects of knowledge and communication in choosing mother-baby care options.

DETAILED DESCRIPTION:
Background:

During early postpartum period, mother-infant proximity is important for breastfeeding success. Rooming-in and separate care are both traditional practices. Rooming-in involves keeping the mother and the baby together in the same room after birth during hospitalization, whereas separate care keeps the baby in the hospital baby room. Using decision aid (DA) is one way to provide information to pregnant women and to involve them in making decisions about their mother-baby care approaches.

Patients and Methods:

Decision aids are interventions designed to help pregnant women to choose their options of mother-baby care by providing information on those options and any potential outcome relevant to different mother-baby care options. Pregnant women considering mother-baby care approaches are randomly assigned to receive a DA or the standard oral information (control condition) during consultation.

By asking the pregnant women to look into a series of paired-comparisons, the DA leads the pregnant women to consider the competing attributes (i.e. specific risks/benefits) of the care options. The primary outcomes are decision conflicts and decision-making difficulties after consultation.

Hypothesis:

The pregnant women of the DAs group are predicted to have lower decisional conflict scores before labor and lower decision regret scores after labor compared with controlled women. Our study hopes to support the efficacy of DAs in helping pregnant women to arrive at mother-care decision.

ELIGIBILITY:
Inclusion Criteria:

Women delivered by cesarean section or induction between 37 weeks, 0 days and 41 weeks, six days.

Exclusion Criteria:

Pregnant women with preeclampsia, mental disorder, do not understand Chinese, and newborn baby with infection, or not suitable for rooming-in care.

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 150 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Decision conflicts | An average of 3 days after delivering
  Total score of decisional conflict scale

SECONDARY OUTCOMES:
Decision regret | An average of 3 days after delivering
  Total score of decision regret

CONTACTS AND LOCATIONS:
Overall Officials: Ka-Wai Tam, MD, PhD, Principal Investigator — No.291, Zhongzheng Rd., Zhonghe , Taipei 23561, Taiwan. Shuanghe Hospital
Locations (1):
- Ka-Wai Tam, New Taipei City, Taiwan